CLINICAL TRIAL: NCT04645667
Title: Development of a Population Pharmacokinetic Model to Optimize Tacrolimus Dosing in Adult Recipients of Allogeneic Hematopoietic Stem Cell Transplant.
Brief Title: Tacrolimus in Allogeneic Hematopoietic Stem Cell Transplant (HCT)
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC2034; IRB 19-3328 (Other: University of North Carolina at Chapel Hill)
Record Dates: First submitted 2020-11-18; First posted 2020-11-27 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Acute GVHD
Keywords: tacrolimus; aGVHD; pharmacokinetics; pharmacodynamics; pharmacogenomics; CYP3A5 genetic polymorphisms
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood will be collected at baseline prior to the first dose of tacrolimus, and will will consist of 2 tubes of 5 mL blood (one for PK and one pharmacogenetics). Then, serial blood sampling will occur at 0.5, 1, 2, 4, 6, and 10h after the first tacrolimus dose. On Day -2 and Day -1, blood will be collected prior to the morning dose for the 24h and 48h estimates. On Day 0, blood will again be collected at 0.5, 1, 2, 4, 6, and 10. Also, 10 mL of blood on Day +1, Day +8, and Day +15 (30 mL total) for PD biomarker analysis. For haplo-transplant patients, blood sampling will be similar but will occur on Day +5, Day +6, Day +7, and Day +8 once tacrolimus is initiated, and blood for PD biomarkers will occur on Day +9, Day +16, and Day +23.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients of allogeneic hematopoietic HCT: Patients who receive their first allogeneic HCT transplant and who receive tacrolimus for aGVHD prophylaxis per standard of care.
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — Patients will be enrolled into this group if they receive tacrolimus per standard of care. This is an observational study and no interventions will be made.
  Other Names: Prograf

SUMMARY:
The purpose of this research study is to evaluate tacrolimus plasma concentrations in patients who will undergo an allogeneic hematopoietic stem cell transplant (HCT). The study aims to identify associations between plasma concentrations, baseline demographic characteristics, clinical lab parameters, and genetic factors. These associations will help clinicians determine the best starting dose for tacrolimus in order to minimize risks of aGVHD and tacrolimus-induced toxicities.

DETAILED DESCRIPTION:
This study aims to evaluate tacrolimus concentration-time data to characterize tacrolimus inter-individual pharmacokinetic (PK) variability in adult patients who will receive HCT, and to associate concentration-time data, exposure and clearance data with important clinical endpoints such as acute graft-versus-host disease (aGVHD) and tacrolimus-induced toxicities. This study proposes to enroll 50 patients at University of North Carolina Medical Center (UNCMC) who will undergo allogeneic HCT, who will receive tacrolimus starting the third day prior to allogeneic HCT (Day -3) for aGVHD prophylaxis. This will be an observational study, and its goal will be to ideally collect baseline clinical and demographic data, concentration-time data for tacrolimus on Day -3 (3 days before the transplant), Day -2 (2 days before the transplant), Day -1 (one day before the transplant), and Day 0 (the day of the allogeneic HCT) for a full pharmacokinetic profile. A medical chart review will be conducted to extract data on tacrolimus-induced toxicities (i.e., acute kidney injury [AKI], hypertension, metabolic panel changes, etc.) and aGVHD incidence rate up to Day +100 (100 days post-allogeneic HCT). Blood will also be collected for genotyping and will also be collected after the transplant to obtain information for surrogate PD biomarkers of tacrolimus efficacy, such as interleukin 2 (IL2) production and quantifiable nuclear localization of the dephosphorylated nuclear-activated T cells (NFAT). These data will aid in the development of a population-based PK/pharmacodynamic (PD) model that will serve as the foundation for a proposed precision dosing approach to optimize tacrolimus dosing. One of the secondary endpoints will be time to aGVHD, which will be defined as the duration from D0 until the first occurrence of aGVHD, censored at 100 days post-allogeneic HCT (Day +100). In the case of haplo-transplant patients, they will receive tacrolimus starting on Day +5 (as opposed to on Day -3 in non-haplo-transplant recipients). Per standard of care, haplo-transplant patients are initiated on Day +5 (5 days after the transplant). Therefore, in these patients, serial blood draws will be collected on a similar timeline as the non-haplo-transplant patients, but in this case Day +5, Day +6 (6 days after the transplant), Day +7 (7 days after the transplant), and Day +8 (8 days after the transplant; Day +8 is when they reach steady-state). For the PD biomarker studies in haplo-transplant patients, blood draws will occur on Day +9 (9 days after the transplant), Day +16 (16 days after the transplant), and Day +23 (23 days after the transplant) (Figure 2). All other procedures will remain the same.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age
2. Patients who will undergo their first HCT
3. Patients who will start tacrolimus for aGVHD prophylaxis
4. Patients who have provided written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization for release of personal health information

Exclusion Criteria:

1. Patients who have cognitive impairments that could affect informed decision-making
2. Patients who are incarcerated
3. Patients started on a strong CYP3A4 inhibitor (i.e. posaconazole)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is a single-center prospective observational study that seeks to characterize steady-state tacrolimus pharmacokinetics pharmacodynamics in adult recipients of their first allogeneic HCT. Adult subjects who receive prophylactic tacrolimus for aGVHD prevention, and who receive active follow-up surveillance at our institution, are eligible for enrollment. The study population will consist of subjects treated in the Inpatient Bone Marrow Transplant Unit at the University of North Carolina Medical Center. A total of 50 subjects will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Tacrolimus clearance | Day +1 of tacrolimus administration to Day +4 of tacrolimus administration
  Patient's clearance calculated after the first day on tacrolimus and patient's clearance calculated after 5-6 doses of tacrolimus after they reach steady-state

SECONDARY OUTCOMES:
Incidence and severity of aGVHD | Day +21 to Day +100 from HCT
  The duration from the day of transplant to the first occurrence of aGVHD, censored at 100 days post-HCT.
Incidence of tacrolimus-induced toxicities | Day -3 to Day +100 from HCT
  The duration from the day of transplant to the first occurrence of tacrolimus-induced toxicities (AKI, hypertension, and metabolic abnormalities)
Time to aGVHD | Day +21 to Day +100 from HCT
  The duration from the day of transplant to the first occurrence of aGVHD, censored at 100 days post-HCT.
Time to tacrolimus-induced toxicities (AKI, hypertension, metabolic panel abnormalities) | Day -3 to Day +100 from HCT
  The duration from the day of transplant to the first occurrence of AKI, hypertension, and metabolic panel abnormalities, censored at 100 days post-HCT.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Crona, PharmD, PhD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mahmoud HK, Elhaddad AM, Fahmy OA, Samra MA, Abdelfattah RM, El-Nahass YH, Fathy GM, Abdelhady MS. Allogeneic hematopoietic stem cell transplantation for non-malignant hematological disorders. J Adv Res. 2015 May;6(3):449-58. doi: 10.1016/j.jare.2014.11.001. Epub 2014 Nov 7. PMID 26257943
- [Background] Broder MS, Quock TP, Chang E, Reddy SR, Agarwal-Hashmi R, Arai S, Villa KF. The Cost of Hematopoietic Stem-Cell Transplantation in the United States. Am Health Drug Benefits. 2017 Oct;10(7):366-374. PMID 29263771
- [Background] Yalniz FF, Murad MH, Lee SJ, Pavletic SZ, Khera N, Shah ND, Hashmi SK. Steroid Refractory Chronic Graft-Versus-Host Disease: Cost-Effectiveness Analysis. Biol Blood Marrow Transplant. 2018 Sep;24(9):1920-1927. doi: 10.1016/j.bbmt.2018.03.008. Epub 2018 Mar 14. PMID 29550629
- [Background] Thomson AW, Bonham CA, Zeevi A. Mode of action of tacrolimus (FK506): molecular and cellular mechanisms. Ther Drug Monit. 1995 Dec;17(6):584-91. doi: 10.1097/00007691-199512000-00007. PMID 8588225
- [Background] Ganetsky A, Shah A, Miano TA, Hwang WT, He J, Loren AW, Hexner EO, Frey NV, Porter DL, Reshef R. Higher tacrolimus concentrations early after transplant reduce the risk of acute GvHD in reduced-intensity allogeneic stem cell transplantation. Bone Marrow Transplant. 2016 Apr;51(4):568-72. doi: 10.1038/bmt.2015.323. Epub 2015 Dec 21. PMID 26691423
- [Background] Kuypers DR, Claes K, Evenepoel P, Maes B, Vanrenterghem Y. Clinical efficacy and toxicity profile of tacrolimus and mycophenolic acid in relation to combined long-term pharmacokinetics in de novo renal allograft recipients. Clin Pharmacol Ther. 2004 May;75(5):434-47. doi: 10.1016/j.clpt.2003.12.009. PMID 15116056
- [Background] Przepiorka D, Devine S, Fay J, Uberti J, Wingard J. Practical considerations in the use of tacrolimus for allogeneic marrow transplantation. Bone Marrow Transplant. 1999 Nov;24(10):1053-6. doi: 10.1038/sj.bmt.1702032. PMID 10578154
- [Background] Staatz CE, Tett SE. Clinical pharmacokinetics and pharmacodynamics of tacrolimus in solid organ transplantation. Clin Pharmacokinet. 2004;43(10):623-53. doi: 10.2165/00003088-200443100-00001. PMID 15244495
- [Background] Birdwell KA, Decker B, Barbarino JM, Peterson JF, Stein CM, Sadee W, Wang D, Vinks AA, He Y, Swen JJ, Leeder JS, van Schaik R, Thummel KE, Klein TE, Caudle KE, MacPhee IA. Clinical Pharmacogenetics Implementation Consortium (CPIC) Guidelines for CYP3A5 Genotype and Tacrolimus Dosing. Clin Pharmacol Ther. 2015 Jul;98(1):19-24. doi: 10.1002/cpt.113. Epub 2015 Jun 3. PMID 25801146
- [Background] Hesselink DA, Bouamar R, Elens L, van Schaik RH, van Gelder T. The role of pharmacogenetics in the disposition of and response to tacrolimus in solid organ transplantation. Clin Pharmacokinet. 2014 Feb;53(2):123-39. doi: 10.1007/s40262-013-0120-3. PMID 24249597
- [Background] Provenzani A, Santeusanio A, Mathis E, Notarbartolo M, Labbozzetta M, Poma P, Provenzani A, Polidori C, Vizzini G, Polidori P, D'Alessandro N. Pharmacogenetic considerations for optimizing tacrolimus dosing in liver and kidney transplant patients. World J Gastroenterol. 2013 Dec 28;19(48):9156-73. doi: 10.3748/wjg.v19.i48.9156. PMID 24409044
- [Background] Astellas Pharma US. Prograf (tacrolimus) [package insert]. U. S. Food and Drug Administra-tion website. https://www.accessdata.fda.gov/drugsatfda_docs/label/2012/050709s031lbl.pdf. Revised May 2018. Accessed Feburary 7, 2020.
- [Background] Bremer S, Vethe NT, Skauby M, Kasbo M, Johansson ED, Midtvedt K, Bergan S. NFAT-regulated cytokine gene expression during tacrolimus therapy early after renal transplantation. Br J Clin Pharmacol. 2017 Nov;83(11):2494-2502. doi: 10.1111/bcp.13367. Epub 2017 Aug 16. PMID 28686294
- [Background] Venkataramanan R, Swaminathan A, Prasad T, Jain A, Zuckerman S, Warty V, McMichael J, Lever J, Burckart G, Starzl T. Clinical pharmacokinetics of tacrolimus. Clin Pharmacokinet. 1995 Dec;29(6):404-30. doi: 10.2165/00003088-199529060-00003. PMID 8787947
- [Background] Undre NA. Pharmacokinetics of tacrolimus-based combination therapies. Nephrol Dial Transplant. 2003 May;18 Suppl 1:i12-5. doi: 10.1093/ndt/gfg1029. PMID 12738758
- [Background] Wallemacq PE, Verbeeck RK. Comparative clinical pharmacokinetics of tacrolimus in paediatric and adult patients. Clin Pharmacokinet. 2001;40(4):283-95. doi: 10.2165/00003088-200140040-00004. PMID 11368293
- [Background] Moller A, Iwasaki K, Kawamura A, Teramura Y, Shiraga T, Hata T, Schafer A, Undre NA. The disposition of 14C-labeled tacrolimus after intravenous and oral administration in healthy human subjects. Drug Metab Dispos. 1999 Jun;27(6):633-6. PMID 10348790
- [Background] Dai Y, Hebert MF, Isoherranen N, Davis CL, Marsh C, Shen DD, Thummel KE. Effect of CYP3A5 polymorphism on tacrolimus metabolic clearance in vitro. Drug Metab Dispos. 2006 May;34(5):836-47. doi: 10.1124/dmd.105.008680. Epub 2006 Feb 24. PMID 16501005
- [Background] Hebert MF. Contributions of hepatic and intestinal metabolism and P-glycoprotein to cyclosporine and tacrolimus oral drug delivery. Adv Drug Deliv Rev. 1997 Sep 15;27(2-3):201-214. doi: 10.1016/s0169-409x(97)00043-4. PMID 10837558
- [Background] Anglicheau D, Verstuyft C, Laurent-Puig P, Becquemont L, Schlageter MH, Cassinat B, Beaune P, Legendre C, Thervet E. Association of the multidrug resistance-1 gene single-nucleotide polymorphisms with the tacrolimus dose requirements in renal transplant recipients. J Am Soc Nephrol. 2003 Jul;14(7):1889-96. doi: 10.1097/01.asn.0000073901.94759.36. PMID 12819250
- [Background] Furlong T, Storb R, Anasetti C, Appelbaum FR, Deeg HJ, Doney K, Martin P, Sullivan K, Witherspoon R, Nash RA. Clinical outcome after conversion to FK 506 (tacrolimus) therapy for acute graft-versus-host disease resistant to cyclosporine or for cyclosporine-associated toxicities. Bone Marrow Transplant. 2000 Nov;26(9):985-91. doi: 10.1038/sj.bmt.1702639. PMID 11100278
- [Background] US Department of Health and Human Services. Common Terminology Criteria for Adverse Events (CTCAE). 5.0. National Institutes of Health; 2017. https://ctep.cancer.gov/protocolDevelopment/electronic_applications/docs/CTCAE_v5_Quick_Reference_5x7.pdf
- [Background] Center for International Blood and Marrow Transplant Research Transplant Activity Report Covering 2010-2014.
- [Derived] Dunlap TC, Zhu J, Weiner DL, Kemper RM, DeVane SC, Ma F, Nguyen V, Coghill JM, Dang V, Grgic T, Jamieson K, Miller J, Myers J, Patel T, Riches M, Serody JS, Trepte M, Vincent BG, Wood WA, Ptachcinski JR, Shaw JR, Weimer E, Armistead PM, Crona DJ. A Tacrolimus Population Pharmacokinetic Model for Adult Allogeneic Hematopoietic Cell Transplant Recipients Provides Clinical Opportunities for Precision Dosing. Clin Pharmacokinet. 2025 Nov;64(11):1621-1637. doi: 10.1007/s40262-025-01529-w. Epub 2025 Aug 12. PMID 40794300
- [Derived] Zhu J, Campagne O, Torrice CD, Flynn G, Miller JA, Patel T, Suzuki O, Ptachcinski JR, Armistead PM, Wiltshire T, Mager DE, Weiner DL, Crona DJ. Evaluation of the performance of a prior tacrolimus population pharmacokinetic kidney transplant model among adult allogeneic hematopoietic stem cell transplant patients. Clin Transl Sci. 2021 May;14(3):908-918. doi: 10.1111/cts.12956. Epub 2021 Jan 27. PMID 33502111